## Clinical evaluation of the effect of the scanning pattern on complete-arch implant scans (strategies IOS)

C.I. 22/645-E

November, 23th, 2022

Informed Consent Form

## INFORMED CONSENT

| I, | (name | of | participant/patient) |
|---|---|---|---|
| | | | , on behalf |
| of myself, and | acknowledging that I | have taken in | nto account your previously |
| expressed wish | nes or objections reg | arding this s | tudy, I confirm that I have |
| read the inform | nation sheet that has b | been delivere | d to me. I affirm that I have |
| understood wh | at it puts in it and th | at I have bee | en given the opportunity to |
| ask the questio | ns that I have conside | ered necessar | y to be able to understand it |
| well, for which | I express my free an | d informed w | vill to voluntarily accept my |
| participation in | the study "Accuracy | and scannin | g time in different full-arch |
| intraoral digita | l impression systems | ", I subscribe | e that a copy of this consent |
| is given to m | e and I expressly | consent, thro | ough my signature, to the |
| processing of r | ny personal data for | the aforemen | tioned purposes, in relation |
| to the manager | nent and execution o | f the research | n project. |

On \_\_\_\_\_\_ of \_\_\_\_ of 20

| Name and surname |
|-----------------------------------------------------------------------|
| Name and surname of the participant/representative of the researcher: |

## RIGHT OF REVOCATION

(In case you want to exercise your right to withdraw your consent)

I (participant/patient name)

On behalf of myself/or (check all that apply)

On behalf of another person whose name I am going to indicate (check all that apply).

Name of whom I represent:

And, acknowledging having taken into account your previously expressed wishes or objections regarding this study.

Name and surname

Name and surname of the participant/representative of the researcher: